CLINICAL TRIAL: NCT00975663
Title: Evaluation of the Interest of Therapeutic Drug Monitoring of Immunosuppressants (Tacrolimus, Mycophenolate Mofetil) Based on Bayesian Estimation During the Three First Years Following Lung Transplantation, in Patients With or Without Cystic Fibrosis
Brief Title: Bayesian Dose Adjustment of Immunosuppressants After Lung Transplantation
Acronym: BASALT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Marie SENGELEN, CHU Limoges
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I07038
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Lung and Heart-lung Transplantation
Keywords: Lung transplantation; heart-lung transplantation; therapeutic drug monitoring; tacrolimus; mycophenolate; immunosuppressant; pharmacokinetics
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Optimized TDM of tacrolimus and MMF dosing
  Interventions: Drug: Tacrolimus and MMF
- 2 (Active Comparator): Current tacrolimus and MMF dosing strategies
  Interventions: Drug: Tacrolimus and MMF

INTERVENTIONS:
Drug: Tacrolimus and MMF — Tacrolimus: daily oral dose divided into 2 doses (morning and evening). MMF: daily dose divided into 2 doses at 12 hour intervals or 3 doses at 8 hour intervals.
  Arms: 1
Drug: Tacrolimus and MMF — Tacrolimus: daily oral dose divided into 2 doses (morning and evening). MMF: daily dose divided into 2 doses at 12 hour intervals or 3 doses at 8 hour intervals.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate in lung or heart-lung transplant patients on tacrolimus and mycophenolate the impact of optimized mofetil (MMF) therapeutic drug monitoring and dose adjustment of both drugs on the incidence of treatment failure over the first three years post-transplantation.

DETAILED DESCRIPTION:
This research will be based on a prospective randomized trial comparing optimized TDM of tacrolimus and MMF to the current strategy of tacrolimus and MMF dose adjustment in lung transplant recipients. The study will focus on the first three years post-transplantation, as treatment failures (including BOS) occur mainly during this post-transplantation period. As the aim of tacrolimus and MMF dose individualization is to avoid over- or underexposure, for the purpose of this study treatment failure will be a composite criterion gathering events which reflect both over- and underexposure to tacrolimus and MMF.

Optimized TDM of tacrolimus and MMF based on blood tacrolimus and plasma MPA AUC Bayesian estimation will be compared to current strategies: tacrolimus dose adjustment based on trough levels (C0) and administration of a standard dose of MMF, decreased by the pulmonologist in case of adverse drug reactions or increased in case of inefficacy. The efficacy of optimized strategy vs. current strategies will be mainly evaluated through the incidence of treatment failure.

ELIGIBILITY:
Inclusion Criteria

* Male and female patients aged 18 years or more
* CF and non-CF patients receiving single-lung or double-lung or heart-lung transplantation for the first time
* Patients on oral tacrolimus and MMF for at least 48 hours at the time of inclusion (administration via a naso-gastric tube possible if necessary)
* Patients without progressive chronic pathology jeopardizing short term patient and graft survival
* Patients accepting to comply with at least the evaluation visits planned in the investigation center over the first three years post-transplantation (D7, D14, M1, M3, M6, M12, M18, M24, M30, M36)
* Patients giving their free and informed written consent to participate in this study
* Patients with a health insurance policy or registered under a health insurance program

Exclusion Criteria:

* Patients aged less than 18 years or patients over 18 years under guardianship
* Patients who disagree with this research
* Patients with a contra-indication to receiving tacrolimus or MMF
* Patients on cyclosporine, sirolimus or everolimus
* Patients who have already benefited from a solid organ transplantation in the past (including lung or heart-lung transplantation)
* Patients infected by Burkholderia cenocepacia (Burkholderia cepacia genomovar III)
* Patients receiving HIV protease inhibitors (major pharmacokinetic interaction with tacrolimus)
* Pregnant or breastfeeding women or those of child-bearing age who do not use an efficient contraceptive method
* Drug users or patients suffering from neuro-psychiatric disorders preventing them from both proper comprehension of the protocol and reliable consent
* Patients already participating in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Immunosuppressive treatment failure | Day 7, day 14, day 21; months 3, 6 and every six months afterwards up to 3 years posttransplantation

SECONDARY OUTCOMES:
Efficacy score | Day 7, day 14, day 21; months 3, 6 and every six months afterwards up to 3 years posttransplantation
Toxicity score | Day 7, day 14, day 21; months 3, 6 and every six months afterwards up to 3 years posttransplantation
Benefit/risk ratio | Day 7, day 14, day 21; months 3, 6 and every six months afterwards up to 3 years posttransplantation
Each event composing the composite criterion | Day 7, day 14, day 21; months 3, 6 and every six months afterwards up to 3 years posttransplantation
Overall cost of patients monitoring | Day 7, day 14, day 21; months 3, 6 and every six months afterwards up to 3 years posttransplantation
Pharmacogenetic and proteomic analysis | Day 7, day 14, day 21; months 3, 6 and every six months afterwards up to 3 years posttransplantation

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MARQUET, MD, Study Director — CHU Limoges
Locations (9):
- Service de Pneumologie, Brussels, Belgium
- France (8):
  - Pôle Médecine Aiguë et Communautaire, Clinique de Pneumologie,, Grenoble
  - Service de Pneumologie, HCL Lyon, Lyon
  - ApHm -Chirurgie thoracique, Marseille
  - Service de Pneumologie-CHU de Nantes, Nantes
  - Service de Chirurgie Cardiovasculaire - Hôpital Georges Pompidou, Paris
  - Service de Pneumologie - CH de Suresnes, Paris
  - Service de Pneumologie - Phtisiologie - Hôpital Bichat, Paris
  - Service de Pneumologie - CHU de Strasbourg, Strasbourg